CLINICAL TRIAL: NCT06709131
Title: A Clinical Study to Investigate the Safety and Efficacy of CT0991 in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: A Clinical Study to Explore the Safety and Efficacy of CT0991 in Relapsed/Refractory Acute Myeloid Leukemia
Acronym: CT0991
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Product manufacturing process improvement
Sponsor: He Huang (Other)
Responsible Party: Sponsor-Investigator, He Huang, Principal Investigator, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2024024
Record Dates: First submitted 2024-11-22; First posted 2024-11-29 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia(AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells（ chimeric antigen receptor T cells） (Experimental): CAR-T cells（ chimeric antigen receptor T cells）
  Interventions: Drug: CAR-T cells（ chimeric antigen receptor T cells）

INTERVENTIONS:
Drug: CAR-T cells（ chimeric antigen receptor T cells） — CAR-T cells（ chimeric antigen receptor T cells）

SUMMARY:
A Clinical Study to Investigate the Safety and Efficacy of CT0991 in Patients with Relapsed/Refractory Acute Myeloid Leukemia

DETAILED DESCRIPTION:
This is a single-arm, open-label, dose-escalation clinical trial to evaluate the safety, efficacy, and cellular pharmacokinetics of CT0991 in patients with relapsed or refractory acute myeloid leukemia. It is planned to enroll 9-24 participants in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the clinical trial; Fully understand and are informed of this study and sign the informed consent form; Willing to follow and able to complete all trial procedures；
2. Age 18-75 years (inclusive), male or female；
3. Estimated survival > 12 weeks;
4. Patients with relapsed or refractory AML as defined in the Chinese Guidelines for the Diagnosis and Treatment of Relapsed and Refractory Acute Myeloid Leukemia (Version 2023);
5. ECOG score 0-2;
6. Participants should meet the following test results (no ongoing ongoing supportive care): a)Left ventricular ejection fraction (LVEF) > 50%; b)ALT ≤ 2.5 × ULN, AST ≤ 2.5 × ULN, total bilirubin ≤ 2 × ULN; c)Endogenous creatinine clearance ≥ 30 mL/min (creatinine clearance calculated using the Cockcroft-Gault formula); d) Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN and prothrombin time (PT) ≤ 1.5 × ULN.
7. Female participants of childbearing potential must have a negative serum pregnancy test at screening and before receiving cleansing, be willing to use a highly effective and reliable method of contraception for 1 year after receiving trial treatment, and be absolutely prohibited from donating eggs for 1 year after receiving trial treatment during the trial;
8. Male participants willing to use a highly effective and reliable method of contraception for 1 year following trial treatment if sexually active with a woman of childbearing potential. All male participants were absolutely prohibited from donating sperm for 1 year after receiving trial treatment during the trial.

Exclusion Criteria:

1. The participant has any serious illness, laboratory abnormality, or psychiatric disorder that may impair the ability to receive or tolerate planned trial treatment; or the investigator judges that the participant 's participation in the clinical trial is not in his/her best interest (e.g., compromised health), or may hinder, limit, or confound protocol-specific assessments;
2. Participants were diagnosed with acute promyelocytic leukemia (APL), BCR-ABL positive leukemia (chronic myeloid leukemia in acute phase), secondary AML (other than MDS), central nervous system leukemia;
3. Participants with a history of epilepsy or other central nervous system disease;
4. Participants who have received autologous stem cell transplantation within 12 weeks or allogeneic stem cell transplantation within 6 months prior to screening;
5. Participant has clinically significant active GVHD or is receiving systemic corticosteroids for GVHD;
6. Participant has a second primary malignancy other than AML that has required treatment or has not been in complete remission within the past 2 years. The following cancers were considered curable, including nonmetastatic basal cell or squamous cell skin cancer, nonmetastatic prostate cancer, breast or cervical carcinoma in situ, and nonmuscle-invasive bladder cancer. Participants receiving ongoing hormonal therapy may be included in this trial at the discretion of the medical monitor in consultation with the investigator;
7. Participants had positive serology for human immunodeficiency virus (HIV) and syphilis, active hepatitis C virus (HCV) infection, or active hepatitis B virus (HBV) infection. Participants with a history of previously treated hepatitis B or C were allowed to be included in this trial if viral load could not be detected by qPCR and/or nucleic acid testing;
8. Major surgery within 14 days prior to washout or planned major surgery within 28 days after receiving CT0991 infusion. If required, the medical monitor and investigator must discuss to confirm whether the surgery is considered a major surgery before the participant is included in this trial;
9. Received anti-tumor therapy 14 days before Preconditioning, including chemotherapy, molecular targeted therapy;
10. Systemic therapeutic doses of glucocorticoids (defined as ≥ 20 mg prednisone or other equivalent per day) within 14 days prior to cleansing; however topical glucocorticoids such as topical dermal, eye drops, nasal sprays, inhalations, and physiologic replacement therapy doses of glucocorticoids are permitted ;
11. Vaccination with live attenuated vaccine or mRNA vaccine within 4 weeks prior to clear shower;
12. Allergic or intolerant to clear shower drugs and tocilizumab, or allergic to DMSO in cell infusion preparations, or previous history of other serious allergies such as anaphylactic shock;
13. Toxicities caused by previous treatment did not recover to Common Terminology Criteria for Adverse Events (CTCAE) ≤ Grade 1, except alopecia, peripheral neuropathy, and other events that were judged by the investigator to be unlikely to be cumulative toxicities due to clear shower or CT0991 infusion;
14. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-08-17 (Actual); Study Completion 2026-08-17 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) after CT0991infusion | 12 months after CT0991 infusion
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria
Dose-limiting toxicity （DLT） | Up to 28 days after CAR-T cells infusion
  The DLT is evaluated as the proportion of patients who experienced adverse events related to CT0991 that meet the criteria for DLT events after the first infusion.
MTD and/or dose range | Up to 28 days after CAR-T cells infusion
  Evaluate Dose limited toxicity and recommended dosage range after CT0991 infusion

SECONDARY OUTCOMES:
Complete response (CR), and complete response with incomplete hematologic recovery (CRi) | 12 months after CT0991 infusion
  Performed according to the Technical Guidelines for Clinical Development of New Drugs for Acute Myeloid Leukemia and ELN 2022 Criteria for AML defined of Achieve CR and CRi.
complete response with partial hematologic recovery (CRh), Morphologic leukemia-free status (MLFS) and partial response (PR) | 12 months after CT0991 infusion
  Performed according to the Technical Guidelines for Clinical Development of New Drugs for Acute Myeloid Leukemia and ELN 2022 Criteria for AML defined of Achieve CRh, MLFS and PR.
Duration of response (DOR) | 12 months after CT0991 infusion
  Participants achieving CR/CRi/CRh will be included in the analysis set for DOR. DOR is defined as the time from the date of confirmed response until the date of disease relapse or death from any cause, whichever occurs first.
Event-free survival (EFS) | 12 months after CT0991 infusion
  defined as the time from the date of receiving the infusion to the date of treatment failure (failure to achieve CR/CRh/CRi/MLFS/PR after both efficacy assessments), or relapse (hematologic relapse or extramedullary relapse after CR/CRh/CRi), or death from any cause, whichever occurs first. When an EFS event was "Ineffective Therapy", the primary analysis of EFS was performed on a 1-day basis (ie, time to treatment received as the event). For a more comprehensive assessment, sensitivity analyses could be performed using the actual date of treatment failure, end of treatment, or start of next-line anti-leukemia therapy as the end of EFS for treatment failure, respectively.
Overall survival (OS) | 12 months after CT0991 infusion
  defined as the time from the date of receiving the infusion to the date of death from any cause.
Minimal Residual Disease (MRD) Negative Rate | 12 months after CT0991 infusion
  tested in all participants who achieved CR/CRh/CRi. MRD negativity was defined as abnormal cells detected by the MFC method accounting for < 0.1% of CD45-positive cells (at least 500,000 CD45-positive cells detected).
Test Copy number of CAR | 12 months after CT0991 infusion
  Evaluate cellular pharmacokinetics of CT0991

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No